CLINICAL TRIAL: NCT00199225
Title: Evaluation of Possible Effects on the QT/ QTc Interval of Rupatadine in Healthy Volunteers: A Randomised, Parallel, Placebo and Positive Controlled Study
Brief Title: Evaluation of Possible Effects on the QT/ QTc Interval of Rupatadine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: J. Uriach and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IC012RUP/1/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-09

CONDITIONS: Human Experimentation (Human Volunteers)
Keywords: Thorough study QT/QTc; Cardiac repolarization; QT prolongation
MeSH Terms: conditions — Long QT Syndrome | interventions — rupatadine; Moxifloxacin

INTERVENTIONS:
Drug: Rupatadine
Drug: moxifloxacin
Procedure: Continous electrocardiographic register
Procedure: Pharmacokinetic profile

SUMMARY:
This phase I trial will evaluate the effects of rupatadine, at a dose of 10 mg OD (authorised and marketed dose) and the 100mg/day (supratherapeutic dose) on the ECG parameters with a special focus on its effect on cardiac repolarisation (QTc interval duration).Furthermore, the study is performed to assess the pharmacokinetic-pharmacodynamic relationship between plasma concentration of rupatadine and its effects, if any, on cardiac repolarisation mainly in the QTc interval).

The main objective is to assess whether administration of a repeated dose of 10 and 100 mg/day , has the potential to cause QT prolongation in healthy volunteers.

DETAILED DESCRIPTION:
Recently, as FDA as EMEA provides recommendations to sponsors concerning the design, conduct, analysis and interpretation of clinical studies to assess the potential for delaying cardiac repolarisation. This paper recommends to perform a 'through Qt/QTc' study to expand ECGs safety evaluation during later stages of drug development. It was recomended that the study was randomized, blind and placebo controlled. Moreover, as a high sensitivy is necessary in order to detect differences in the QTc measure, it was essential a positive control included. On that basis, the positive control should be well-characterized and consistently produce an effect corresponding to the largest change in the QT/QTc interval that is currently viewed as clinically not important to detect (a mean change of around 5 ms. Because of this, we decide select as positive control: moxifloxacin, used in the most of similar phase I clinical trials.

In these type of studies, as recommended by the guidelines, there should be a caracterization to ensure that the dose-response and generally the concentration-response relationship for QT/QTc prolongation, including exploration of concentrations that are higher than those achieved following the therapeutic doses. So, thererfore, we decided use 100 mg/daY (10 times the therapeutic dose) as supratherapeutic dose to be administered.

We decide propose a new phase I study as recommended guidelines (a single-blind, randomised, placebo and active-controlled, parallel design). With this, we've tried complet the rupatadine effects over QTc and another electrocardiographic parameters and valued the risk-benefit relationship for this new antiH1 and PAF antagonist

single

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for admission to the study:

1. Male or female between 18 and 45 years old (inclusive)
2. In good health as determined by the principal investigator based on medical history, physical examination, ECG, and clinical laboratory tests
3. Body Mass Index between 19 and 27 kg/m2.
4. Non-smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication)
5. Negative serology Hepatitis B, C or HIV in the 3 previous months
6. Female subjects must have a negative serum pregnancy test result prior to enrollment into the study. Female subjects of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must be using appropriate birth control (defined as a method which results in a low failure rate, i.e. less than 1% per year, when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices [IUDs], sexual abstinence, or a vasectomised partner) during the entire duration of the study. Oral contraceptive medications are prohibited in this study
7. Capable of understanding and complying with the protocol and must have signed the informed consent document prior to performance of any study-related procedures

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Currently abusing drugs or alcohol (> 30 gr/day; or > 1/2 drinks/day for females/males, defined according to USDA Dietary Guidelines 2000) or with a history of drug or alcohol abuse within the past two years
2. Subjects will be asked to consume xanthine-containing food and beverages (eg, coffee, tea, chocolate, and cola beverages).
3. Has taken any grapefruit or grapefruit juice during 14 days prior the screening visit and day -1.
4. Unwilling or unable to comply with the protocol or reside in the study unit during the study period or to cooperate fully with the principal investigator and site personnel
5. Has used any prescription medication within 14 days prior to Day 0, or over-the-counter (OTC) medication, herbal preparations, and/or vitamins within 48 hours prior to the start of study drug administration on Day 0
6. A 12 lead ECG obtained at screening with: PR > 240 msec, QRS >110 msec and QTc > 430 msec in males or QTc > 430 msec in females, bradycardia (<50 lpm) or clinically significant minor STT wave changes on the screening ECG, or any other changes on the screening ECG that would interfere with measurement of the QT interval
7. Has a serum potassium, sodium, calcium, or magnesium level that is not within normal limits or has other laboratory values outside the normal range at the screening visit that are deemed by the principal investigator to make the subject an inappropriate candidate for the study
8. Has taken any other investigational drug during the 2 months prior to screening visit
9. Has donated or lost more than a unit of blood within 30 days prior to screening visit
10. Has any condition(s) that in the investigator's opinion would: a) warrant exclusion from the study or b) prevent the subject from completing the study
11. Unable to understand verbal and/or written the informed consent.
12. History of hypersensitivity or allergic reaction to moxifloxacin or any other member of the quinolone class of antibiotics
13. History of hypersensitivity or allergic reaction to rupatadine or any other antihistamine compounds

Furthermore, will be excluded during the study all the subjects that shows any waiver to the inclusion or exclusion criteria, under the criteria of principal investigator and/or medical monitor.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160
Dates: Start 2005-02; Study Completion 2005-07

PRIMARY OUTCOMES:
To assess whether administration of a repeated dose of 10 and 100 mg/day , has the potential to cause QT prolongation in healthy volunteers, according the current guidelines.

SECONDARY OUTCOMES:
Furthermore, the study is performed to assess the pharmacokinetic-pharmacodynamic relationship between plasma concentration of rupatadine and its effects, if any, on cardiac repolarisation mainly in the QTc interval).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Barbanoj, MD, Principal Investigator — Institut de Recerca-Hospital de la Santa Creu i Sant Pau; Rosa Mª Antonijoan, MD, Principal Investigator — Institut de Recerca- Hospital de la Santa Creu i Sant Pau; Esther G Donado, PhD, Study Director — J. Uriach and Company; Iñaki Izquierdo, MD, Study Chair — J. Uriach and Company
Locations (1):
- Centre de Investigació de Medicaments-Intitut de Recerca-Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain